CLINICAL TRIAL: NCT04574596
Title: MDRO: Study of Highly Resistant Escherichia Coli
Brief Title: Multi-Drug Resistant Organism (MDRO): Study of Highly Resistant Escherichia Coli
Acronym: SHREC
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00106280; UM1AI104681 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-10-05 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2020-09

CONDITIONS: E Coli Infection
Keywords: Extended Spectrum β-Lactamases (ESBL)
MeSH Terms: conditions — Escherichia coli Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3GCRceftriaxone-resistant-E. coli in blood culture
  Control group 3GCSceftriaxone-susceptible-E. coli in a blood culture :
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3GCR ceftriaxone-resistant-E. coli: Positive blood culture for above resistant e coli. Observational there will be no intervention
  Interventions: Other: no Intervention
- 3GCS ceftriaxone-susceptible-E. coli: Positive blood culture for above susceptible e coli. Observational there will be no intervention
  Interventions: Other: no Intervention

INTERVENTIONS:
Other: no Intervention — This is an observational study. There is no intervention

SUMMARY:
This is a prospective, observational, multicenter, case-control study.

DETAILED DESCRIPTION:
This is an observational cohort study. A total of 300 subjects will be enrolled. Cases are defined as unique subjects who have a monomicrobial blood culture positive for growth of 3rd Generation Cephalosporin Resistant Escherichia coli (3GCR-Ec), defined as resistance to ceftriaxone or cefotaxime, during hospitalization. For each case, the next available unique subject from the same study site, with a monomicrobial blood culture positive for growth of 3rd Generation Cephalosporin Sensitive Escherichia coli (3GCS-Ec) during hospitalization will be included as a control. A waiver of informed consent and HIPAA will be requested. This is a minimal risk study without any direct subject contact. In addition, no subject information will be collected that is not part of routine clinical care.

The trigger for enrollment in the study will be the identification in a participating local microbiology laboratory of a 3GCR-Ec in a monomicrobial blood culture. These will be reported to study personnel at the study site, who will evaluate eligibility. If the subject is deemed eligible, the 3GCR-Ec isolate will be saved for shipping to the Laboratory Center, and the isolate also saved at the local laboratory. Sites will be advised to destroy any samples saved at the local laboratory as part of this study at the end of the study. The local microbiology laboratory, or designee, will then identify the next subject available with a 3GCS-Ec in a blood culture. These will also be reported to study personnel for evaluation of eligibility as a control. If the control subject is eligible, the corresponding 3GCS-Ec isolate will be saved for shipping to the Laboratory Center, and the isolate will also be saved at the local laboratory . Sites will be advised to destroy any samples saved at the local laboratory as part of this study at the end of the study.

For cases and controls, clinical data will be collected from the electronic health records (EHR) for up to 30 days after the index blood culture. Data collection will be performed by study personnel at the site into a central, secure, research database.

One E. coli isolate per study subject will be collected from the index blood culture. No other biologic samples will be collected. Data will be entered at or after the 30-day time point. There will be no long-term follow-up for subjects.

Primary Objective:

To evaluate the use of oral step down therapy in subjects with 3GCR-Ec and 3GCS-Ec bacteremia.

Secondary Objectives

1. To describe the treatment regimens used in subjects with 3GCR-Ec and 3GCS-Ec bacteremia.
2. To determine the association between duration of intravenous antibiotics and Inverse Probability Weighting (IPW)-adjusted Desirability Of Outcome Ranking (DOOR) outcomes at 30 days
3. To determine the association between total duration of antibiotics and IPW-adjusted DOOR outcomes at 30 days
4. To determine risk factors on days 0, 3, 5, and 7 after first positive blood culture for poor outcomes (either DOOR composite score or individual outcomes) at 30 days.

Exploratory Objective:

• To describe phenotypic and genotypic characteristics of bacterial isolates.

This study is minimal risk to study participants, and has no data safety monitoring board.

ELIGIBILITY:
Inclusion criteria:

1. Positive monomicrobial blood culture for 3GCR-Ec (cases) or 3GCS-Ec (control)
2. Hospitalized at the time of obtaining index blood culture OR in the emergency department at the time of obtaining index blood culture, if followed by hospitalization within 72 hours

Exclusion criteria:

1. Previously included in this study as either control or case subject
2. Previous blood culture positive for E. coli during the current hospitalization
3. In vitro non-susceptibility to any carbapenem tested in the local clinical microbiology laboratory
4. Evidence of carbapenemase production in the E. coli isolate of interest as determined by the local clinical microbiology laboratory

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Sample size: 300 total: 150 3GCR-Ec cases, 150 3GCS-Ec controls.
  * This is a consecutive cohort study without age or gender exclusions. Special populations such as women, children, and minorities will be included.
  * The study population will be drawn from subjects who are hospitalized at participating study hospitals.
  * This observational study is minimal-risk and will be performed under a waiver of consent and HIPAA.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who received oral step-down therapy | Within 30 days of culture collection
  Number of participants who received oral-step down therapy for treatment of e. Coli

SECONDARY OUTCOMES:
Duration of antibiotics | From culture collection to 30 days post culture collection
  Total duration of antibiotics
Duration of intravenous antibiotics | From culture collection to 30 days post culture collection
  Total duration of intravenous antibiotics
Duration of oral antibiotics | From culture collection to 30 days post culture collection
  Total duration of oral antibiotics
Number of participants who received short course antibiotic therapy | From culture collection to 30 days post culture collection
  Number of participants who received short-course antibiotic therapy defined as <= 7 days of antibiotic therapy
Number of participants with ongoing antibiotic treatment at 30 days | 30 days post culture collection
  Number of participants with ongoing antibiotic treatment at 30 days
Number of participants with resolution or improvement of symptoms | 30 days post culture collection
  Number of participants with resolution or improvement of symptoms by 30 days
Number of participants with anatomic source specific symptomatic response | 30 days post culture collection
  Number of participants with anatomic source specific symptomatic response
Discharged by 30 days | culture collection through 30 days post culture collection
  Discharged from the hospital by 30 days
Days to discharge | culture collection through 30 days post culture collection
  Days from culture collection to hospital discharge
Length of stay | hospital admission through 30 days post culture collection
  Days from hospital admission to hospital discharge
Number of participants with a readmission within 30 days of index culture | culture collection through 30 days post culture collection
  Number of participants with a readmission to the same hospital within 30 days of index culture
Number of participants with a new positive blood culture with E. coli within 30 days of index culture | culture collection through 30 days post culture collection
  Number of participants with a new positive blood culture with E. coli within 30 days of index culture
Number of participants with a three-fold or greater increase in serum creatinine from day of index culture | culture collection through 30 days post culture collection
  Number of participants with a three-fold or greater increase in serum creatinine from day of index culture
Number of participants with a newly required renal replacement therapy post index culture | culture collection through 30 days post culture collection
  Number of participants with a newly required renal replacement therapy post index culture
Number of participants with a Clostridioides difficile infection | culture collection through 30 days post culture collection
  Number of participants with a Clostridioides difficile infection
Mortality at 30 days | culture collection through 30 days post culture collection
  Mortality at 30 days
Number of participants in the ICU on day 0, 3, 5, and 7 | Days 0, 3, 5, 7
  Number of participants in the ICU on day 0, 3, 5, and 7
Desireability of Outcome Ranking (DOOR) outcome at 30 days | 30 days post culture collection
  The desirability of outcome ranking (DOOR) in this study will assess three deleterious events (lack of clinical response, unsuccessful discharge, and undesirable events) in addition to survival at 30 days after the index culture. The five ordered levels of the variable, from best to worst, are:
  1. Alive without deleterious events
  2. Alive with 1 deleterious event
  3. Alive with 2 deleterious events
  4. Alive with 3 deleterious events
  5. Death by 30 days
  The undesirable events are:
  * Post-culture renal failure
  * Clostridioides difficile infection

OTHER OUTCOMES:
Antibiotic resistance phenotype | Day 0, which is the date of culture collection in this observational study
  Antibiotic resistance phenotype
Antimicrobial resistance genes | Day 0, which is the date of culture collection in this observational study
  Antimicrobial resistance genes
Duration of individual antibiotics and specific combinations of antibiotics | culture collection through 30 days post culture collection
  Duration of individual antibiotics and specific combinations of antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Vance G. Fowler, MD, Study Director — Duke Clinical Research Institute; David van Duin, MD, PhD, Principal Investigator — University of North Carolina
Locations (13):
- United States (13):
  - Harbor-University of California Los Angeles Medical Center, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Ochsner Medical Center, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical College, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No